CLINICAL TRIAL: NCT06850337
Title: Characterization of Megakaryocytic Subpopulations and the "Immune" Phenotype of Platelets of the Sickle Cell Disease Patient
Brief Title: Megakaryocyte Heterogeneity in Sickle Cell Disease
Acronym: MegaDrep
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH2_2024/04; 2024-A01093-44 (Other: ANSM)
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: sickle cell disease; immune megakaryocytes; platelets; CD48; CD148
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A specific research sample corresponding to a 5 ml tube of blood and a 5 ml tube of bone marrow (only for orthopedic surgery patients) will be taken during the inclusion visit for sickle cell patients.
  For patients without sickle cell , after verification of the eligibility criteria and collection of their agreement to participate, a 5 ml blood tube will be taken with determination of their AA genotype (on hemoglobin electrophoresis). As well as the collection of a 5 ml blood tube and a 5 ml bone marrow tube will be taken following the surgical procedure. Once the AA genetic status is confirmed, the bone marrow sample will be processed. Otherwise, the sample will be destroyed and the patient will not be included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- SS patients: patients with SS sickle cell disease
- SC patients: patients with SC sickle cell disease
- control group AA: patient without sickle cell disease (AA hemoglobin)

SUMMARY:
Sickle cell disease (SCD) is characterized by chronic hemolytic anemia, painful crisis called vaso-occlusive crisis (VOC) and chronic inflammation. Activated platelets of SCD patients participated to both chronic inflammation and painful VOC. Platelets are anucleated cells from the fragmentation of megakaryocytes in bone marrow.

The main aim of this study is to characterize the distribution of the different megakaryocyte subpopulations of sickle cell disease patients SS and SC and in particular the "immune" megakaryocytes CD148+CD48+ and to compare it with the platelet phenotype.

DETAILED DESCRIPTION:
Platelets are activated in all sickle cell disease patients at baseline with higher expression of selective P (CD62P). Platelets provide a major function in primary hemostasis by the formation of the platelet clot and also participate in coagulation through the formation of an electro-negative phospholipid surface essential to the enzymes of the coagulation cascade. It is now known that platelets are also immune cells that are able to secrete pro-inflammatory cytokines (TGF beta, IFN gamma), that they express certain Toll-like receptors (TLR4) and the inflammasome NLRP3 leading to the activation of caspase-1. Several teams, including ours, have shown that inflammasome and/or caspase-1 can be activated in an infectious context, particularly viral (dengue fever, COVID) and inflammatory (chronic inflammatory bowel diseases, etc.).

Platelets are anucleated cells from the fragmentation of megakaryocytes. Their protein profile is therefore the result of bone marrow differentiation of megakaryocytes. Recently, it has been shown a cellular heterogeneity within megakaryocytes including immune megakaryocytes whose proportion can significantly increase in stress and inflammation condition. It is not clear whether these immune megakaryocytes that could behave as antigen-presenting cells are capable of producing blood platelets.

We wonder whether sickle cell disease patients have a different proportion of these immune megakaryocytes compared to healthy subjects and whether their activated blood platelets carry specific markers of these immune megakaryocytes.

SCD patients will be recruited in the active file of the sickle cell center of Guadeloupe. Two groups of patients will be constituted: SS patients and SC patients. The control group will be composed of patients who come for hip or knee replacement and do not suffer from chronic disease. Only one blood and bone marrow collection will be realized during the study.

ELIGIBILITY:
Inclusion Criteria:

* patients with SS or SC SCD
* diagnosis of SCD performed by electrophoresis or HPLC in a reference laboratory for hemoglobinopathies
* patients older than 18 years at inclusion
* clinically in a steady state at inclusion (without complication in the last month and without transfusion in the three last months)
* patient followed up for SCD at the sickle cell center of Guadeloupe (University hospital of Guadeloupe, Pointe à Pitre)
* patients who will provide written informed consent in accordance with the Declaration of Helsinki
* patients affiliated to national social security
* the control group (AA subjects) will be patients older than 18 years old who come at the University hospital of Guadeloupe, (Pointe à Pitre) for hip or knee replacement and will do not suffer from chronic disease.

Exclusion Criteria:

* patients younger than 18 years old
* patients with hemoglobinopathy other than SS and SC SCD
* patients with a transfusion therapy or on bleeding therapy for less than three months
* patients no affiliated to national social security
* pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with sockle celle disease are patients who come for their disease. Control group are patients who come at the University hospital of Guadeloupe (Pointe à Pitre), for hip or knee replacement and will do not suffer from chronic disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
proportion of immune megakaryocytes CD148+CD48+ in bone marrow | 24 months
  The primary outcome will be the evaluation of the proportion of immune megakaryocytes CD148+CD48+ in bone marrow of sickle cell disease patients in comparison to control group.

SECONDARY OUTCOMES:
platelet phenotype | 24 months
  The secondary outcomes are to compare the platelet phenotype between the three groups of patients, including the proportion of CD148+CD48+ platelets, to study the activation of this platelet subpopulation (expression of CD62P) and establish whether there is a relationship between the proportion of immune megakaryocytes in the bone marrow and the proportion of CD148+CD48+ platelets in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Baccini, MD PhD, Study Chair — CHU de la Guadeloupe
Locations (1):
- Chu de La Guadeloupe, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No